CLINICAL TRIAL: NCT02347371
Title: Follow-up Registry of Heart Transplant Recipients, to Determine Long Term Outcome and Need for Further Interventional and Non-interventional Procedures
Brief Title: Heart Transplant Registry of Városmajor
Status: Completed | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: VSZR - 001
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Disorder Related to Cardiac Transplantation
Keywords: Heart transplant; Cardiac allograft vasculopathy; Chronic rejection; Immunosuppressant therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to determine the long term outcomes of heart transplantations performed at the Semmelweis University Heart and Vascular Center. All eventual interventional and non-interventional procedures will be accounted for and summarized.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant recipient
* >18 years old
* Signed informed consent
* Cared for at the Semmelweis University Heart and Vascular Center

Exclusion Criteria:

* Denies consent to registry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant recipient, cared for by the Semmelweis University Heart and Vascular Center
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Outcome of heart transplantation as measured by all-cause mortality | 5 years
  All-cause mortality will be assessed after transplantation in all participating subjects.

SECONDARY OUTCOMES:
Morbidity after heart transplantation | 5 years
  All invasive procedures that are required after initial surgery will be tracked and accounted for.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Merkely, MD PhD DSc, Principal Investigator — Semmelweis University Heart and Vascular Center
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, Hungary